CLINICAL TRIAL: NCT03090672
Title: Use of Cellular and Biocellular Therapy in Musculoskeletal Pain, Dysfunction, Degenerative or Inflammatory Disease
Brief Title: Cellular & Biocellular Regenerative Therapy in Musculoskeletal Pain, Dysfunction,Degenerative or Inflammatory Disease
Acronym: BRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Robert W Alexander, MD (Other)
Collaborators: Regeneris Medical (Other); Global Alliance for Regenerative Medicine (Other)
Responsible Party: Sponsor-Investigator, Robert W Alexander, MD, Principal Investigator, Regeneris Medical
Organization: Regeneris Medical (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGV MSK 1
Record Dates: First submitted 2017-03-06; First posted 2017-03-27 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis; Rheumatoid Nodule; Degenerative Joint Disease; Tendinopathy; Tendinosis; Back Pain
Keywords: Arthritis; Degenerative; Tendinosis; Jont disease; Low back pain
MeSH Terms: conditions — Osteoarthritis; Rheumatoid Nodule; Joint Diseases; Tendinopathy; Back Pain; Arthritis; Low Back Pain | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tSVF + PRP Arm1 (Experimental): Stromal Vascular Fraction tSVF + Platelet Rich Plasma (PRP) concentrate
  Interventions: Procedure: Tissue Stromal Vascular Fraction; Biological: Platelet Rich Plasma
- tSVF + PRP + cSVF Enrichment Arm 2 (Experimental): tissue Stromal Vascular Fraction (tSVF) + Platelet-Rich Plasma (PRP) concentration + (cSVF)
  Interventions: Procedure: Tissue Stromal Vascular Fraction; Biological: Platelet Rich Plasma; Procedure: Cellular Stromal Vascular Fraction
- Normal Saline IV + cSVF Arm 3 (Experimental): Cellular Stromal Vascular Fraction (cSVF); Normal Saline IV introduction
  Interventions: Drug: Normal Saline; Procedure: Cellular Stromal Vascular Fraction

INTERVENTIONS:
Drug: Normal Saline — Normal Saline IV delivery
  Arms: Normal Saline IV + cSVF Arm 3
Procedure: Tissue Stromal Vascular Fraction — tSVF
  Arms: tSVF + PRP + cSVF Enrichment Arm 2; tSVF + PRP Arm1
Biological: Platelet Rich Plasma — PRP
  Arms: tSVF + PRP + cSVF Enrichment Arm 2; tSVF + PRP Arm1
Procedure: Cellular Stromal Vascular Fraction — cSVF
  Arms: Normal Saline IV + cSVF Arm 3; tSVF + PRP + cSVF Enrichment Arm 2

SUMMARY:
Musculoskeletal disorders and degeneration represent injuries or pain in the body's joint ligaments, tendons, muscles, nerves, and skeletal elements that support extremities, spine and related tissues. Direct injuries and aging contribute to breakdown and inflammation of these tissues, leading to debilitation and loss of function in these areas. This has major impact on quality of life, occupational/recreation limitations, and psychosocial implications.

Many therapies have been employed including medications, physical therapy, occupational therapy, and a variety of surgical interventions each of which have distinct limitations, often covering the issues versus providing actual healing and return to function. Many reports are now available utilizing self-healing options which include use of stem/stromal cellular therapy or biocellular treatments (either from adipose or marrow) using targeted placement of cells, matrix and platelet concentrates. Termed cellular or Biocellular therapy (typically optimized using ultrasound guidance). It is proposed that use of cellular isolates or cell-stroma derived from the largest deposit of these cells (adipose greater than marrow), may use in conjunction with targeted placement or as a stand alone methodology intravascular use.

This study is designed as a interventional means to examine the safety and efficacy of the use of cellular and tissue stromal vascular fraction in musculoskeletal pain, dysfunction degeneration or inflammatory disorders.

DETAILED DESCRIPTION:
Musculoskeletal disorders and degeneration represent injuries or pain in the body's joint ligaments, tendons, muscles, nerves, and skeletal elements that support extremities, spine and related tissues. Direct injuries and aging contribute to breakdown and inflammation of these tissues, leading to debilitation and loss of function in these areas. This has major impact on quality of life, occupational/recreation limitations, and psychosocial implications.

Many therapies have been employed including medications, physical therapy, occupational therapy, and a variety of surgical interventions each of which have distinct limitations, often covering the issues versus providing actual healing and return to function. Many reports are now available utilizing self-healing options which include use of stem/stromal cells (either from adipose or marrow) using targeted placement of cells, matrix and platelet concentrates. This is termed Biocellular therapy, and typically is optimized by use of ultrasound guidance. It is proposed that use of cellular isolates derived from the largest deposit of these cells (adipose greater than marrow), may use in conjunction with targeted placement or as a stand alone methodology of parenteral use.

This study is designed as a interventional means to examine the safety and efficacy of the use of cellular stromal vascular fraction (cSVF) in musculoskeletal pain, dysfunction degeneration or inflammatory disorders. The important cellular components represent, not the adipocyte, but the heterogeneous cell group associated with the peri-vasculature. The group does include certain cells referred to as "stem" or "stromal" cells, and are considered key elements of cellular and biocellular treatments. The carrier microvascular tissue, adipose, has been shown to not participate in wound healing or cellular replacement per se. It is well established that those perivascular (adventitial) cell types are found in essentially all tissues of the body, but in highest numbers in the easily accessed depots with the subdermal fat. It is proposed that areas of these groups are responded to as a result of "signaling" to permit a chemotactic request for needed growth factors and cytokines which effectively contribute to the healing capability at failing or damaged sites. This Trial will investigate the safety/efficacy of either combining specific targeting (ultrasound) with and/or without systemic parenteral route introduction.

This study includes closed syringe, disposable microcannula harvesting of subdermal fat tissues for obtaining the native perivascular stromal elements (extracellular matrix (ECM) and periadventitial cells shown to be multipotent (in potentials), incubation, digestion and isolation of cSVF. This isolated and concentration of stem/stromal cellular pellet (without actual extracellular matrix or stromal scaffolding elements) is then suspended in 500 cc sterile Normal Saline (NS) and deployed via peripheral intravenous route. Evaluations of safety issues are measured at intervals (both severe and non-severe categories) and by ultrasound and imaging studies.

Biocellular treatments are defined as use of tissue stromal vascular fraction (tSVF) obtained within adipose tissue complex (ATC), combined with high density platelet rich plasma (HD PRP) concentrated from standard blood draw. Concentration in FDA approved platelet concentrate devices to achieve levels of >4 times patient's own measured baseline levels. Such concentrates have been shown to provide important growth factors and cytokines (signal proteins) naturally involved in wound healing and repair functions. A form of Cell-Enriched Biocellular Therapy (CEBT) is available as a component of this study, in which the tSVF + HD PRP can be enhanced in cellular numbers via the process of isolating and concentrating cSVF discussed above. Many small case series and case reports have been published in the peer reviewed medical literature which suggest that these interventions are both safe and effective at relieving musculoskeletal disorders included in the study.

This study in intended to provide evidence of a non-drug safety and efficacy using both of these interventions. Evaluation and tracking of adverse events or severe adverse events (SAE) will be tracked according to intervals described. Examination of the optimal numbers of cells, viability of such cells, and evaluation of the efficacy will be statistically studied reported relative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented inflammatory, autoimmune (rheumatoid arthritis (RA), degeneration of musculoskeletal system
* No systemic disorders which, in the opinion of the principal investigators or provider, would disqualify from being safely able to undergo needed procedures
* Able to provide informed consent
* Patient having adequate donor adipose (fat) tissue
* Patient mature enough to tolerate the needed procedures

Exclusion Criteria:

* Systemic or psychological impairment which would preclude patient tolerance and understanding of procedures and follow up
* Patients with known active cancer and chemotherapy or radiation therapy
* Patients with ongoing active infections
* High dose steroid users or use of injections of corticoid steroids within a six month timeframe
* Opiate addition or in treatment program for withdrawal
* History of severe traumatic brain injuries
* If, in the opinion of providers, the patient will not be able to fully cooperate or complete the study and its follow up

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-03-11 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants with complications | 1 month
  Adverse and Severe Adverse Events Reports

SECONDARY OUTCOMES:
Change from baseline quality of life level (QoL Questionnaire) | 6 months, 12 months
  QoL Questionnaire
Change from baseline visual analog pain score | 6 months, 1 year, 2 year
  Changes of Visual Analog Pain Score (VAS) 1-10
Change from baseline of limitation of activities (Functional analysis of range of motion) | baseline, 6 months, 1 year
  Functional analysis of range of motion compared from baseline
Change from baseline of imaging if required for study entry | baseline, 1 year
  imaging

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Alexander, MD, Principal Investigator — GARM USA; Glenn C Terry, MD, Principal Investigator — Global Alliance for Regenerative Medicine (GARM); Ryan JP Welter, MD, PhD, Principal Investigator — Regeneris Medical
Locations (1):
- Regeneris Medical, North Attleboro, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Comparative analysis of safety and efficacy between use of ultrasound guided tissue stromal vascular fraction (AD-tSVF) plus high density platelet rich plasma (HD-PRP) with use of intravascular deployment of adipose-derived cellular stromal vascular fraction (AD-cSVF)

REFERENCES:
- [Background] Kuorinka I, Jonsson B, Kilbom A, Vinterberg H, Biering-Sorensen F, Andersson G, Jorgensen K. Standardised Nordic questionnaires for the analysis of musculoskeletal symptoms. Appl Ergon. 1987 Sep;18(3):233-7. doi: 10.1016/0003-6870(87)90010-x. PMID 15676628
- [Background] Gallagher S, Heberger JR. Examining the interaction of force and repetition on musculoskeletal disorder risk: a systematic literature review. Hum Factors. 2013 Feb;55(1):108-24. doi: 10.1177/0018720812449648. PMID 23516797
- [Background] Alexander, Robert W., Understanding Mechanical Emulsification (NanoFat) Versus Enzymatic Isolation fo Tissue Stromal Vascular Fraction (tSVF) From Adipose Tissue: Potential Uses in Biocellular Regenerative Medicine. J of Prolo. 2016; 8: 3947-960.
- [Background] Alexander RW. Biocellular Regenerative Medicine: Use of Adipose-Derived Stem/Stromal Cells and It's Native Bioactive Matrix. Phys Med Rehabil Clin N Am. 2016 Nov;27(4):871-891. doi: 10.1016/j.pmr.2016.06.005. PMID 27788905
- [Background] Alderman, D, Alexander, R.W.,: Advances In Regenerative Medicine: High Density Platelet-Rich Plasma and Stem Cell Prolotherapy. J Pract Pain Management, 2011; Vol Oct: 49-90
- [Background] Alexander, Robert W., Understanding Adipose-Derived Stromal Vascular Fraction (SVF) Cell Biology On The Basis of Perivascular Cell Components In Aesthetic and Regenerative Medicine. J. Prolo; 2012; 4: e13777
- [Background] Alexander RW, Harrell DB. Autologous fat grafting: use of closed syringe microcannula system for enhanced autologous structural grafting. Clin Cosmet Investig Dermatol. 2013 Apr 8;6:91-102. doi: 10.2147/CCID.S40575. Print 2013. PMID 23630430
- [Background] Nelson AE, Allen KD, Golightly YM, Goode AP, Jordan JM. A systematic review of recommendations and guidelines for the management of osteoarthritis: The chronic osteoarthritis management initiative of the U.S. bone and joint initiative. Semin Arthritis Rheum. 2014 Jun;43(6):701-12. doi: 10.1016/j.semarthrit.2013.11.012. Epub 2013 Dec 4. PMID 24387819
- [Background] Katz JN, Brownlee SA, Jones MH. The role of arthroscopy in the management of knee osteoarthritis. Best Pract Res Clin Rheumatol. 2014 Feb;28(1):143-56. doi: 10.1016/j.berh.2014.01.008. PMID 24792949
- [Background] Thorlund JB, Juhl CB, Roos EM, Lohmander LS. Arthroscopic surgery for degenerative knee: systematic review and meta-analysis of benefits and harms. BMJ. 2015 Jun 16;350:h2747. doi: 10.1136/bmj.h2747. PMID 26080045
- [Background] Burdett N, McNeil JD. Difficulties with assessing the benefit of glucosamine sulphate as a treatment for osteoarthritis. Int J Evid Based Healthc. 2012 Sep;10(3):222-6. doi: 10.1111/j.1744-1609.2012.00279.x. PMID 22925619
- [Result] Oliver, K., Alexander, RW. Combination of Autologous Adipose-Derived Tissue Stromal Vascular Fraction Plus High Density Platelet-Rich Plasma or Bone Marrow Concentrates in Achilles Tendon Tears. J. Prolo; 2013; 5: e895-912.